CLINICAL TRIAL: NCT06921083
Title: Investigating Management and Perceptions of Aggression, Conflict, and Threat in ICU Environments
Brief Title: Violence in ICU: Outcomes, Lessons, and Experiences of ICU Team (The VIOLENT-Study)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2024-01621; am25Sutter2
Record Dates: First submitted 2025-03-20; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Workplace Stress
Keywords: Intensive Care Unit; Workplace Violence
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the perceptions, experiences, and responses of healthcare professionals working in intensive care units in Switzerland concerning patient violence.

DETAILED DESCRIPTION:
Workplace violence, as defined by the International Labor Organization, includes any action, incident, or behavior that assaults, threatens, harms, or injures a person during their work. Healthcare workers face the highest risk of workplace violence among all professions. Violence can take many forms, including verbal abuse, physical offenses to sexual harassment. While most research focuses on psychiatric and emergency departments, workplace violence in intensive care units (ICUs) is understudied and often underreported. As a result, little is known about its prevalence and risk factors, leading to a lack of awareness and effective prevention strategies.

This study examines the perceptions, experiences, and responses of healthcare professionals in Swiss ICUs. A questionnaire-based survey will assess various aspects, including personal background (such as education and professional role), the frequency and nature of past incidents of workplace violence, responses and measures taken, psychological or professional consequences, current prevention strategies, and suggestions for improving workplace safety.

Since workplace violence is a common issue, the results of this study could help improve the work environment and safety in ICUs and other healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Consenting nurses and physicians currently working in Swiss intensive care units
* Nurses and physicians consenting to participate will be included

Exclusion Criteria:

* Nurses and physicians who do not consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nurses and physicians working in the intensive care unit at Swiss hospitals
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demographic information (ICU Staff Questionnaire) | 2025
  Participants provide demographic details, including gender and age, using a questionnaire.
Completion date (ICU Staff Questionnaire) | 2025
  The date of questionnaire completion is recorded.
Professional background (ICU Staff Questionnaire) | 2025
  Assessment of professional role of the intensive care unit (ICU) staff, including their education and work experience, using a questionnaire.
Frequency of violent incident (ICU Staff Questionnaire) | 2025
  Participants report the frequency of violent incidents encountered from patients or their relatives in the ICU setting, using a questionnaire.
Type of violent incident (ICU Staff Questionnaire) | 2025
  Participants report the type of violent incidents (verbal, physical, and sexual) encountered from patients or their relatives in the ICU setting, using a questionnaire.
Characteristics of violent incident (ICU Staff Questionnaire) | 2025
  Participants provide detailed information about specific violent incidents they have experienced in the ICU, including the context and perceived triggers, using a questionnaire.
Reporting of violent incident (ICU Staff Questionnaire) | 2025
  Participants report whether the violent incident has been reported, using a questionnaire.
Personal impact of workplace violence (ICU Staff Questionnaire) | 2025
  Participants describe the personal impact of workplace violence, including psychological and mental health consequences, using a questionnaire.
Professional impact of workplace violence (ICU Staff Questionnaire) | 2025
  Participants report how workplace violence influences professional factors such as job satisfaction and workload, using a questionnaire.
Actions taken during or after violent incident (ICU Staff Questionnaire) | 2025
  Participants report the responses and measures taken during or after the violent incident, using a questionnaire.
Strategies for enhancing workplace safety in the ICU (ICU Staff Questionnaire) | 2025
  Participants provide information on strategies for enhancing workplace safety in the ICU, such as existing institutional policies, prior training in handling workplace violence, and their opinions on workplace violence prevention and recommendations for enhancing ICU safety, using a questionnaire.
Open-ended feedback from participant (ICU Staff Questionnaire) | 2025
  Participants have the opportunity to share additional comments or remarks related to workplace violence and safety in the ICU, using a questionnaire. This information is collected through a freetext field in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Acute Medicine, Intensive Care Unit
Locations (1):
- University Hospital Basel, Intensive Care Unit, Basel, Canton of Basel-City, Switzerland